CLINICAL TRIAL: NCT05864079
Title: Serum Levels of Developmental Endothelial Locus-1 and Its Relationship With Platelet Count and Soluble P-selectin in Overweight and Obese Subjects
Brief Title: Developmental Endothelial Locus-1, Platelet Count, and Soluble P-selectin in Overweight and Obese Subjects
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Abdel-mageed Muhammed, Lecturer, Aswan University Hospital
Other Study IDs: DEL-1 and sP-sel in obesity
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: 22 healthy age-matched normal-weight male subjects (BMI is from 18.5 to < 25)
  Interventions: Diagnostic Test: Platelet count; Diagnostic Test: Developmental endothelial locus-1 (DEL-1); Diagnostic Test: soluble P-selectin (sP-sel)
- Overweight: 22 healthy overweight male subjects (BMI is from 25 to < 30). Patients with cardiovascular diseases, any malignancy, hepatic or renal failure, diabetic, hyperthyroid patients, patients with a previous history of thromboembolic diseases, or with a history of major surgery within 60 days will be excluded.
  Interventions: Diagnostic Test: Platelet count; Diagnostic Test: Developmental endothelial locus-1 (DEL-1); Diagnostic Test: soluble P-selectin (sP-sel)
- Obesity: 22 healthy obese male subjects (BMI is ≥ 30). Patients with cardiovascular diseases, any malignancy, hepatic or renal failure, diabetic, hyperthyroid patients, patients with a previous history of thromboembolic diseases, or with a history of major surgery within 60 days will be excluded.
  Interventions: Diagnostic Test: Platelet count; Diagnostic Test: Developmental endothelial locus-1 (DEL-1); Diagnostic Test: soluble P-selectin (sP-sel)

INTERVENTIONS:
Diagnostic Test: Platelet count — Platelet count in study groups
Diagnostic Test: Developmental endothelial locus-1 (DEL-1) — Serum DEL-1 in study groups
Diagnostic Test: soluble P-selectin (sP-sel) — Serum sP-sel in study groups

SUMMARY:
This observational study aims to detect serum levels of Developmental Endothelial Locus-1 (DEL-1), Platelet Count, and Soluble P-selectin (sP-sel) in Overweight and Obese Subjects. The main questions it aims to answer are:

* Is there a difference in serum DEl-1 levels in overweight and obese subjects compared to normal subjects?
* Are there any relations between serum DEL-1 levels, sP-sel, and platelet count in overweight and obese subjects ?

ELIGIBILITY:
Inclusion Criteria:

* Male patients.
* Age (18-65) years.
* Healthy overweight and subjects.

Exclusion Criteria:

* Patients with cardiovascular diseases.
* Diabetic patients.
* Previous history of thrombo-embolic diseases.
* Patients with hyperthyroidism.
* Patients with any type of malignancy.
* Underlying hepatic or renal failure.
* Major surgery within 60 days.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy overweight and obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Platelet count | 6 months
  platelet count in venous blood samples in normal-weight, overweight, and obese subjects
Serum Developmental endothelial locus-1 levels | 6 months
  Serum developmental endothelial locus-1 in normal-weight, overweight, and obese subjects
Serum Soluble P-selectin levels | 6 months
  Serum Soluble P-selectin in normal-weight, overweight, and obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdelmageed Muhammed, lecturer, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hajishengallis G, Chavakis T. DEL-1-Regulated Immune Plasticity and Inflammatory Disorders. Trends Mol Med. 2019 May;25(5):444-459. doi: 10.1016/j.molmed.2019.02.010. Epub 2019 Mar 15. PMID 30885428
- [Background] Purdy JC, Shatzel JJ. The hematologic consequences of obesity. Eur J Haematol. 2021 Mar;106(3):306-319. doi: 10.1111/ejh.13560. Epub 2020 Dec 13. PMID 33270290
- [Background] Barale C, Russo I. Influence of Cardiometabolic Risk Factors on Platelet Function. Int J Mol Sci. 2020 Jan 17;21(2):623. doi: 10.3390/ijms21020623. PMID 31963572
- [Background] Kwon CH, Sun JL, Kim MJ, Abd El-Aty AM, Jeong JH, Jung TW. Clinically confirmed DEL-1 as a myokine attenuates lipid-induced inflammation and insulin resistance in 3T3-L1 adipocytes via AMPK/HO-1- pathway. Adipocyte. 2020 Dec;9(1):576-586. doi: 10.1080/21623945.2020.1823140. PMID 32954935